CLINICAL TRIAL: NCT06238830
Title: Evaluation of Multimodal Analgesia With NOL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-23-4785
Record Dates: First submitted 2024-01-17; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Pain, Postoperative; Analgesia
Keywords: multimodal analgesia; nociceptive level index; NOL; External Oblique Intercostal Plane Block; EIOB
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP M: In patients undergoing elective Laparoscopic Cholecystectomy Surgery, after routine anesthesia induction, a magnesium loading dose of 30 mg/kg will be administered intravenously. Subsequently, a magnesium infusion will be initiated at a rate of 10 mg/kg/hour. Afterward, in the supine position, necessary field preparation and ultrasound (USG) setup will be conducted to administer the External Oblique Intercostal Plane (EOIP) block.The procedure will be applied unilaterally. After desufflation, patients will receive 50 mg dexketoprofen as standard analgesia administered intravenously as a non-steroidal anti-inflammatory drug (NSAID).
- GROUP K: As part of standard analgesia, 50 mg dexketoprofen, administered intravenously as a non-steroidal anti-inflammatory drug (NSAID), will be applied, and these patients will be considered as the control group.
  All patients will undergo general anesthesia induction with 1 µg/kg fentanyl, 2-3 mg/kg propofol, and 0.6 mg/kg rocuronium bromide. During anesthesia maintenance, a mixture of 50% O2 and air will be administered, and sevoflurane will be used at a minimum alveolar concentration of 0.8 (with a target MAC value of 0.8-1.2). Additionally, remifentanil will be administered at a rate of 0.01-0.2 mcg/kg/min. The remifentanil dose range will be increased if the patient's Nociceptive Level (NOL) value remains elevated for 2 minutes when it exceeds 25. BIS monitoring will be performed for all patients, and the BIS value will be maintained between 40-50.

SUMMARY:
The study will include 80 patients undergoing Laparoscopic Cholecystectomy Surgery as part of elective requirements. The study is a single-center, prospective, randomized controlled trial

The aim of the study is

1. To investigate the effectiveness of multimodal analgesia, which includes the newly introduced external oblique intercostal plane block, with the assistance of NOL (Nociception Level), in the management of postoperative pain following commonly performed Laparoscopic Cholecystectomy surgeries.
2. This approach is intended to objectively assess changes in postoperative recovery scores

Patients will be divided into two groups: the Multimodal Analgesia group (Group M), where Erector Obliq Interfascial Plane (EOIP) block, NSAID, and magnesium infusion will be administered, and the control group (Group K).

DETAILED DESCRIPTION:
In the elective laparoscopic cholecystectomy procedures to be performed in the general surgery operating room for 80 patients, 80 envelopes containing written papers indicating the Multimodal Analgesia group (Group M) and the control group (Group K) will be prepared. On the morning of the operation, an envelope will be randomly drawn by operating room personnel in a blinded manner to determine the patient's inclusion group. The patients will be randomized into two groups: the Multimodal Analgesia group (Group M), receiving Erector Oliq Interfascial Plane (EOIP) block, NSAID, and magnesium infusion, and the control group (Group K).

Patients will be informed about the procedures to be performed before the surgery, and written consent will be obtained. After patients are taken to the operating table, standard ASA monitoring (electrocardiogram, non-invasive blood pressure, O2 saturation, body temperature) along with NOL (Nociception Level) and BIS (Bispectral Index) monitoring will be applied. A peripheral venous line will be established on the dorsum of the hand for normal saline infusion. All blocks will be performed under ultrasound guidance.

In Group M, after routine anesthesia induction, intravenous magnesium loading of 30 mg/kg will be followed by an infusion of 10 mg/kg/hour. Subsequently, in the supine position, after the necessary field preparation and ultrasound (USG) setup, a linear ultrasound probe will be positioned sagittally between the mid-clavicular and anterior axillary lines at the level of the 6th rib, with the orientation marker pointing cranially. Identification of the 6th rib can be achieved in two ways: either by placing the ultrasound probe at the level of the lower costal margin where the 10th rib is located and then counting upwards, or by identifying the 7th rib at the level of the xiphoid process and then moving the ultrasound probe one rib upward.

The ultrasound probe will then be rotated to obtain a paramedian sagittal oblique view, with the cranial end slightly medial and the caudal end lateral, approximately 1 to 2 cm medial to the anterior axillary line. Sequentially, from superficial to deep, the following structures will be identified: skin, subcutaneous tissue, external oblique muscle, intercostal muscles between the ribs, pleura, and lung.

For the injection, the skin entry point will be at the medial edge of the anterior axillary line, just cranial to the 6th rib level, using a peripherally directed block needle (Echoplex+, VygonTM, France) advanced in a superomedial to inferolateral plane along the external oblique muscle. The tip of the peripherally directed block needle will be adjusted to the tissue plane between the external oblique and intercostal muscles at the caudal end of the 6th rib and 6th-7th intercostal space. A sterile preparation of 20 mL 0.25% Bupivacaine will be injected into the tissue plane between the 6th and 7th ribs using the hydrodissection technique, and then the peripherally directed block needle will be directed caudally towards the eighth rib.

Using the 'in-plane' method parallel to the ultrasound probe, a negative aspiration will be performed, and a total of 20 mL 0.25% bupivacaine will be injected. The distribution of local anesthetic (LA) will be monitored with ultrasound during the injection. The procedure will be applied unilaterally. Post-desufflation, patients will receive 50 mg dexketoprofen intravenously as standard analgesia.

In Group K, 50 mg dexketoprofen intravenous NSAID will be administered as standard analgesia, serving as the control group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 65 years old
* Those undergoing elective laparoscopic cholecystectomy
* Patients with ASA risk scores of I and II
* Body Mass Index (BMI) < 35 kg/m2
* Patients who have provided informed consent before the procedure
* Individuals who are literate and capable of giving consent.

Exclusion Criteria:

* Patients under 18 years of age and those over 65 years of age
* Individuals with an ASA score of III or higher
* Cases with a surgical duration of less than 60 minutes
* Emergency surgeries
* Those with a history of abdominal surgery
* Pregnant or lactating patients
* Individuals with coagulopathy or using anticoagulant medications
* Those allergic to local anesthetics
* Individuals with localized infection at the injection site
* Patients without the ability to use Patient Controlled Analgesia (PCA) and assess Visual Analog Scale (VAS)
* Patients with peripheral nerve disease
* Individuals with kidney failure and congestive heart failure
* Patients undergoing elective Laparoscopic Cholecystectomy (LK) due to malignancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective laparoscopic cholecystectomy.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Multimodal Analgesia on the Nociceptive Level İndex(NOL) | during surgery time
  The NOL index is a single number between 0 and 100. A NOL between 0 and 25 represents a physiologically suppressed response adequately inhibiting harmful stimuli, indicating sufficient analgesia. A NOL index greater than 25 (continuous or fluctuating) for multiple minutes signifies the patient is perceiving pain. Higher values indicate a stronger nociceptive response. An index consistently below 10 for more than a minute may suggest excessive anti-nociception, prompting consideration for reducing analgesics. If regional analgesia is employed, lower NOL values are anticipated.
  The dosage of remifentanil will be increased if the patient's NOL value remains elevated for 2 minutes when it surpasses 25.The number of changes in Ultiva dosage, NOL values will be recorded before intubation, after intubation, during thoracic entry, and during inflation and deflation, as well as at the time of extubation.

SECONDARY OUTCOMES:
Change From Baseline in Postoperative Recovery Scores on the Visual Analog Scale at Postoperative 30 Minutes | postoperative 30 minute
  The patients will be admitted to the postoperative recovery room. Modified Aldrete scores, PACU discharge, and opioid requirements during this period will be assessed based on postoperative awakening Visual Analog Scale (VAS) values at 0 minutes, 15 minutes, and 30 minutes, considering a value of between 0-10 for VAS. As part of the standard analgesia protocol, patients will receive perioperative 50 mg dexketoprofen. During the postoperative period, VAS monitoring will be conducted, and when VAS values exceed 4, a rescue analgesic of 50 mg tramadol intravenously will be administered and recorded as additional analgesic need.
The intensity of nausea and vomiting | postoperative 30 minute
  Starting from the postoperative recovery room, nausea and vomiting will be assessed. The intensity of nausea and vomiting will be recorded using the following scoring system:
  0: None
  1. Nausea
  2. Retching
  3. Vomiting

CONTACTS AND LOCATIONS:
Overall Officials: AYÇA TUBA DUMANLI ÖZCAN, Principal Investigator — ANKARA BİLKENT CİTY HOSPİTAL

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Kehlet, H., et al., A procedure-specific systematic review and consensus recommendations for postoperative analgesia following laparoscopic cholecystectomy. Surg Endosc, 2005. 19(10): p. 1396-415. — https://link.springer.com/article/10.1007/s00464-004-2173-8
- See also: Tulgar, S., O. Selvi, and M.S. Kapakli, Erector Spinae Plane Block for Different Laparoscopic Abdominal Surgeries: Case Series. Case Rep Anesthesiol, 2018. 2018: p. 3947281. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5835299/